CLINICAL TRIAL: NCT00431210
Title: A Pilot Feasibility Study of Epstein-Barr Virus-Specific Immunotherapy for Nasopharyngeal Carcinoma
Brief Title: Epstein-Barr Virus-Specific Immunotherapy for Nasopharyngeal Carcinoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Jochen Lorch, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-179
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: NPC; EPV
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Biological/Vaccine (Experimental): Epstein-Barr virus-specific adoptive T-cells immunotherapy given intravenously on Days 1 and 14
  Interventions: Biological: Epstein-Barr virus-specific adoptive T-cells immunotherapy

INTERVENTIONS:
Biological: Epstein-Barr virus-specific adoptive T-cells immunotherapy — Given intravenously on Day 1 and Day 14

SUMMARY:
The purpose of this study is to determine the safety of making and giving Epstein-Barr virus (EBV) immunotherapy products to subjects with nasopharyngeal carcinoma (NPC) associated with EBV that has come back or spread to other parts of the body. EBV immunotherapy product is made with white blood cells from the participants body that are collected intravenously. This EBV immunotherapy product may stop cancer cells from growing abnormally. EBV immunotherapy products have been used in several research studies for NPC. Information from these studies suggests the EBV immunotherapy products may stop the growth of NPC in some subjects.

DETAILED DESCRIPTION:
* The first step in this research study is the peripheral blood collection. Approximately 60-90cc's will be collected intravenously and used to prepare the EBV immunotherapy product. It takes about 12 weeks to make the EBV immunotherapy product. During this time, the participant will receive standard of care as prescribed by their doctor.
* The EBV immunotherapy product will be made at a laboratory at the Connell & O'Reilly Families Cell and Manipulation Core Facility at the Dana-Farber Cancer Institute. The EBV immunotherapy product will contain T-cells that may react against your EBV-related tumor.
* A small amount of the EBV product will be used for research studies that will investigate components of the immune system that might be important in effective immunotherapy for NPC.
* EBV immunotherapy product will be given to the participant intravenously (infusion) on the first day of the research study. Fourteen days later, the participant will receive infusion #2. After infusion #2, the research doctor will do some tests to determine the effects that the EBV immunotherapy product has had on the tumor. If the research doctor thinks the participant will benefit from a third infusion then they may receive one.
* Before each infusion of EBV immunotherapy product, a physical examination and blood tests will be performed. During the active treatment phase of this research study, a physical exam and blood tests will be done every 1-2 weeks.
* Before each infusion of EBV immunotherapy product, the research doctor may do a fiberoptic exam of the participants nasopharynx by using a flexible scop to visualize the tumor.
* At 8 weeks post-infusion, we will evaluate the tumor by using a CT scan and/or MRI. We will also perform a PET or PET/CT scan if the research doctor feels it is necessary. We may do a chest CT scan to see if the tumor has spread to the lungs and an abdominal/pelvic CT scan or MRI if the participant has symptoms that suggesting that there may be tumor in the liver, or a bone scan to see if there is tumor in the bones.
* In addition to this study, the research doctor may ask permission to participate in optional research studies. We would like the participants permission to take a biopsy of the tumor after they have received infusion #2. The biopsy will be done by a surgeon who will review the risks of the procedure.
* The participant will return to the clinic for a follow-up visit where the response of the tumor will be evaluated, blood tests and a physical exam will be performed at the following intervals: for the first 2 months after the final infusion, every 2-4 weeks; for month 4 to month 12 after the final infusion, every 2 months; for the second year after the final infusion, every 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically proven NPC of any WHO grade, associated with EBV documented by the presence of EBER by in situ hybridization in the tumor. This must be confirmed by pathology review at Brigham and Women's Hospital.
* Incurable NPC as defined by: relapsed or progressive disease after initial treatment with no potentially curative option; NPC with metastasis
* Recovery from toxicity from any prior NPC therapy to grade 1 or better (CTCACE v.3.0)
* 18 years of age or older
* Evaluable disease, according to RECIST
* ECOG performance status of 0-1
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* Radiotherapy for primary NPC within 8 weeks of enrollment, or radiotherapy for any other reason within 6 weeks
* Chemotherapy for NPC within 2 weeks of enrollment
* Other cancer in the past 5 years, except for carcinoma in situ of the cervix or bladder, or non-melanomatous skin cancer
* Uncontrolled central nervous system metastases
* Acute hepatitis, known HIV, or other condition that requires immunosuppressive therapy, including current use of systemic corticosteroids
* Autoimmune disease that is active and requires current therapy
* Active, uncontrolled, serious infection
* Incomplete healing from previous major surgery
* Significant history of uncontrolled cardiac disease
* Women who have a positive B-hCG test or are breastfeeding
* Any concurrent chemotherapy or other concurrent investigational agent not part of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-02; Primary Completion 2015-06-30 (Actual); Study Completion 2016-01-26 (Actual)

PRIMARY OUTCOMES:
The feasibility and safety of generating and administrating and EBV-specific adoptive T cell in participants with incurable locoregional relapsed and/or distant metastatic EBV-associated NPC. | 2 years

SECONDARY OUTCOMES:
The ability to collect specimens and measure potential biologic correlate of response to therapy | 2 years
time to progression in this patient population | 2 years
median duration of response and median overall survival in this cohort of participants. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Lorch, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
There are no plans to share IPD. Cumulative results will be posted and published.